CLINICAL TRIAL: NCT04124445
Title: Pulsed vs Continuous Radiofrequency Neurotomy for Cervical Facet Joint Mediated Pain: a Single-blind Randomized Controlled Clinical Trial
Brief Title: Pulsed vs Continuous Radiofrequency Neurotomy for Cervical Facet Joint Mediated Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Allevio Pain Management Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16327-16:325610-06-2019
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Faceto-genic Neck Pain; Shoulder Pain Chronic; Faceto-genic Headache
Keywords: Faceto-genic Cervical pain; Chronic pain; Pulsed Radiofrequency ablation; Continues Radiofrequency ablation; Medial Brunch Block
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: After performing patient's eligibility for neck RF and receiving information about procedure, patients will be book for two MBB 4-6 weeks apart. If the patient was eligible after the second MBB, Patient will be asked to sign Informed consent before screening. Screening and recruitment, and randomization, patients will be scheduled for one of the RF techniques.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Radiofrequency Ablation (Active Comparator): Radiofrequency ablation of sensory nerves at minimum 3 levels of cervical spine with Maximum allowable temperature 50° rotation: 90.; Pulse rate: 3 Hz; pulse duration: 50 ms; 3 minutes
  Interventions: Procedure: Pulsed Radiofrequency Ablation
- Continuous Radiofrequency Ablation (Active Comparator): Radiofrequency ablation of sensory nerves at minimum 3 levels of cervical spine, burn will be made at 80° for 60 seconds.
  Interventions: Procedure: Pulsed Radiofrequency Ablation

INTERVENTIONS:
Procedure: Pulsed Radiofrequency Ablation — Radiofrequency ablation, also called rhizotomy, is a nonsurgical, minimally invasive procedure that uses heat to reduce or stop the transmission of pain. Radiofrequency waves ablate, or "burn," the nerve that is causing the pain, essentially eliminating the transmission of pain signals to the brain.
  Other Names: Continuous Radiofrequency Ablation

SUMMARY:
Different studies have revealed different success rates and patient satisfaction after cervical facet C-RF. In a study on 32 patients, with 15 months follow up, 25% had complete pain relief (8). Another study had shown mean pain relief of 12.5 months and 11.5 months following a repeat procedure, with an effectiveness of 95% in 47 patients (8). In one study a success rate of 88% after first RF, and 86% following a repeat RF in 49 patients with facet mediated cervicogenic headache. They regarded the absence of anesthesia in the distribution of the 3rd occipital nerve, a technical failure (9). In a study from New Zealand, demonstrated cervical facet RF as the sole treatment modality, produced 61% -74% complete pain relief with a median duration of 15-17 months in patients who had responded to facet joints diagnostic block (10).

One more study in 2012 has demonstrated high voltage P-RF had a higher short-term effect compare to usual voltage, but results are still lower than C-RF (11). A double blind randomized prospective study has illustrated P-RF did not show any success rate in 6 months pain control, whereas C-RF had 95% pain control for trigeminal neuralgia (12).

Cohen in a recent study has compared P-RF with steroid injection for occipital neuralgia or migraine with occipital nerve tenderness (13). Six weeks pain relief was 61% in P-RF group, and 36% in steroid injection group, with a positive outcome of 34%, and 26% respectively (13). One study on 2010 had reached to 52.6%, 6 months pain improvement on occipital neuralgia (14).

DETAILED DESCRIPTION:
Patients fulfilling eligibility criteria will be randomly allocated to PRF or CRF in a 1:1 ratio. The statistician will use RedCap software to generate random numbers. Patients will be registered to Redcap software and will be concealed from both patients and health care staff. The study coordinator will enter patients' consent and study eligibility information to the Redcap. Once eligible, the Redcap will assign the patient to one of the study group. Patients will be blinded in the proposed study. The assessor is the person who will assess treatment success at the end of the study based on data from completed questionnaires. Questionnaires will be completed every three months by patients through RedCap System. A therapist is the person who will perform the procedure (pain specialist physician). The therapist will not be blinded, because of the nature of intervention.

Patient recruitment is estimated to be completed within 15-24 months. If the required sample size (calculated below) is recruited prior to this time, patient recruitment will be curtailed.

During the first visit the investigator will perform eligibility for neck RF and patient will be received information about the study.

Patients will be book for two MBB 4-6 weeks apart. If the patient was eligible after the second MBB, Patient will be asked to sign Informed consent before screening. Screening and recruitment, and randomization, and administer questionnaires will be performed by research co-ordinator. Study informed consent form (ICF) can be signed on the RF procedure day. If additional visits will be required to finalize the procedures related to the first visit they will be scheduled accordingly. After randomization the qualified participants will be scheduled for their RF.

For the female subjects between the age of 18-50 a pregnancy test will be asked to obtain on screening visit in order to reduce the risk of pregnancy and potential harm to fetus, unless you had previous tubal ligation, or hysterectomy. Post menopause patients are excluded.

Participants will be asked to complete the follow-up questionnaires at 1, 3, 6, 9, and 12 months.

LANSS questionnaire will be asked to be completed 6 weeks after RF. If the score was 12 or higher, patient will be asked to complete them every 4 weeks after till the score reduce to less than 12. LANSS will be sent to the subjects through RedCap software.

On their last study visit, participants will have an exit interview, in addition to completing study measures.

ELIGIBILITY:
Inclusion Criteria:

Age 18-90;

Pain duration > 3 months

Cervical, Shoulder pain or cevicogenic Headache per Pain Diagram;

Two single blinded facet medial branch blocks (MBB) performed 30 days prior to the facet RF;

Subjects show 50% and more pain relief after each MBB (using VAS for this assessment);

Unsuccessful or poorly tolerated previous treatments including: pain control medications, chiropractic, osteopathy, massage therapy, physiotherapy, acupuncture, aqua therapy, Botox injection, and trigger point injection;

Exclusion Criteria:

Non-English speakers;

Refusal to sign informed consent;

Less than 50% pain relief after MBB (using VAS);

Variation in the dose of concomitant pain control medication less than 4 weeks before the procedure;

Allergy to medication or radiology contrast;

Patients with coagulation issues, those currently using anticoagulants and didn't stop them based on Allevio clinic's policy for anticoagulants;

Pregnant patients;

Any pain interventions including previous RF, MBB, infusions 90 days prior to the first MBB for the same area (Except failed Botox injection, and trigger point injection);

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life measurement: Visual Analogue Scale | Beginning of the study , and every 3 months up to 12 months
  Changes in Visual Analogue Scale (VAS), between minimum of zero and maximum of ten
Quality of life measurement: Neck Disability Index | Beginning of the study , and every 3 months up to 12 months
  Changes in the Neck Disability Index - AAOS(NDI_AAOS)
Quality of life measurement: Short Form Brief Pain Inventory | Beginning of the study , and every 3 months up to 12 months
  Changes in the Short Form Brief Pain Inventory (SF-BPI), between minimum of zero and maximum of ten

SECONDARY OUTCOMES:
At least 30% Changes in Pain Score | Beginning of the study , and every 3 months up to 12 months
  Proportion of subjects who achieve at least a 30% decrease in the pain score measured by Visual analogue Scale , between minimum of zero and maximum of ten
At least 30% Changes in Pain Score | Beginning of the study , and every 3 months up to 12 months
  Proportion of subjects who achieve at least a 30% decrease in the pain score measured by Short Form Brief Pain Inventory , between minimum of zero and maximum of ten
At least 30% Changes in Pain Score | Beginning of the study , and every 3 months up to 12 months
  Proportion of subjects who achieve at least a 30% decrease in the pain score measured by The Neck Disability Index , between minimum of zero and maximum of ten
At least 50% Changes in Pain Score | Beginning of the study , and every 3 months up to 12 months
  Proportion of subjects who achieve at least a 50% decrease in the pain score measured by The Neck Disability Index
At least 50% Changes in Pain Score | Beginning of the study , and every 3 months up to 12 months
  Proportion of subjects who achieve at least a 50% decrease in the pain score measured by Short Form Brief Pain Inventory , between minimum of zero and maximum of ten
At least 50% Changes in Pain Score | Beginning of the study , and every 3 months up to 12 months
  Proportion of subjects who achieve at least a 50% decrease in the pain score measured by Visual analogue Scale , between minimum of zero and maximum of ten
Changes in Changes in Global Improvement and Satisfaction | Beginning of the study , and every 3 months up to 12 months
  Changes in Global Improvement and Satisfaction score measured by PGIC
Changes in The Neck Disability Index | Beginning of the study , and every 3 months up to 12 months
  Changes in The Neck Disability Index - AAOS(NDI_AAOS)
Changes in General Anxiety Disorder Questionnaire | Beginning of the study , and every 3 months up to 12 months
  Changes in General Anxiety Disorder Questionnaire (GAD)
Changes in Beck's Depression Inventory | Beginning of the study , and every 3 months up to 12 months
  Changes in Beck's Depression Inventory (BDI)
Changes in Changes in Patients self-reported perceived duration of effect | Beginning of the study , and every 3 months up to 12 months
  Changes in Patients self-reported perceived duration of effect (PSPDE)
Adverse events | Beginning of the study , and every 3 months up to 12 months
  Safety, assessed by the number, severity and duration of adverse reactions. It will be collected as self-rated health-related complaints by the subject and then confirmed medically. The causality will be assigned by the investigator
Pain Medications | Beginning of the study , and every 3 months up to 12 months
  Changes in pain medication use, if it is narcotic, measured by Morphine Equivalent Dose
Changes in Leeds assessment of neuropathic symptoms and signs | 6 weeks after RF and if the score was 12 or higher repeat monthly up to 12 weeks
  Changes in the Leeds assessment of neuropathic symptoms and signs (LANSS), between minimum of zero and maximum of twenty four

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Allevio Pain Management Clinic, Toronto, Ontario
  - Allevio Pain Management, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Results will be published

REFERENCES:
- [Background] Cohen J. Statistical power analysis for the behavioral sciences. 2nd ed. Hillsdale, NJ: L. Erlbaum, 1988.
- [Result] Falco FJ, Erhart S, Wargo BW, Bryce DA, Atluri S, Datta S, Hayek SM. Systematic review of diagnostic utility and therapeutic effectiveness of cervical facet joint interventions. Pain Physician. 2009 Mar-Apr;12(2):323-44. PMID 19305483
- [Result] Yin W, Bogduk N. The nature of neck pain in a private pain clinic in the United States. Pain Med. 2008 Mar;9(2):196-203. doi: 10.1111/j.1526-4637.2007.00369.x. PMID 18298702
- [Result] Gil Faclier, Joseph Kay. Cervical facet radiofrequency neurotomy. Techniques in Regional Anesthesia and Pain Management Volume 4, Issue 3, July 2000, Pages 120-125
- [Result] Smith AD, Jull G, Schneider G, Frizzell B, Hooper RA, Sterling M. Cervical radiofrequency neurotomy reduces central hyperexcitability and improves neck movement in individuals with chronic whiplash. Pain Med. 2014 Jan;15(1):128-41. doi: 10.1111/pme.12262. Epub 2013 Oct 18. PMID 24138594
- [Result] Bogduk N, Govind J. Cervicogenic headache: an assessment of the evidence on clinical diagnosis, invasive tests, and treatment. Lancet Neurol. 2009 Oct;8(10):959-68. doi: 10.1016/S1474-4422(09)70209-1. PMID 19747657
- [Result] Chang MC. Effect of bipolar pulsed radiofrequency on refractory chronic cervical radicular pain: A report of two cases. Medicine (Baltimore). 2017 Apr;96(15):e6604. doi: 10.1097/MD.0000000000006604. PMID 28403104
- [Result] Gazelka HM, Knievel S, Mauck WD, Moeschler SM, Pingree MJ, Rho RH, Lamer TJ. Incidence of neuropathic pain after radiofrequency denervation of the third occipital nerve. J Pain Res. 2014 Apr 10;7:195-8. doi: 10.2147/JPR.S60925. eCollection 2014. PMID 24748815
- [Result] Husted DS, Orton D, Schofferman J, Kine G. Effectiveness of repeated radiofrequency neurotomy for cervical facet joint pain. J Spinal Disord Tech. 2008 Aug;21(6):406-8. doi: 10.1097/BSD.0b013e318158971f. PMID 18679094
- [Result] Govind J, King W, Bailey B, Bogduk N. Radiofrequency neurotomy for the treatment of third occipital headache. J Neurol Neurosurg Psychiatry. 2003 Jan;74(1):88-93. doi: 10.1136/jnnp.74.1.88. PMID 12486273
- [Result] MacVicar J, Borowczyk JM, MacVicar AM, Loughnan BM, Bogduk N. Cervical medial branch radiofrequency neurotomy in New Zealand. Pain Med. 2012 May;13(5):647-54. doi: 10.1111/j.1526-4637.2012.01351.x. Epub 2012 Mar 28. PMID 22458772
- [Result] Fang L, Tao W, Jingjing L, Nan J. Comparison of High-voltage- with Standard-voltage Pulsed Radiofrequency of Gasserian Ganglion in the Treatment of Idiopathic Trigeminal Neuralgia. Pain Pract. 2015 Sep;15(7):595-603. doi: 10.1111/papr.12227. Epub 2014 Jun 23. PMID 24954016
- [Result] Erdine S, Ozyalcin NS, Cimen A, Celik M, Talu GK, Disci R. Comparison of pulsed radiofrequency with conventional radiofrequency in the treatment of idiopathic trigeminal neuralgia. Eur J Pain. 2007 Apr;11(3):309-13. doi: 10.1016/j.ejpain.2006.04.001. Epub 2006 Jun 9. PMID 16762570
- [Result] Cohen SP, Peterlin BL, Fulton L, Neely ET, Kurihara C, Gupta A, Mali J, Fu DC, Jacobs MB, Plunkett AR, Verdun AJ, Stojanovic MP, Hanling S, Constantinescu O, White RL, McLean BC, Pasquina PF, Zhao Z. Randomized, double-blind, comparative-effectiveness study comparing pulsed radiofrequency to steroid injections for occipital neuralgia or migraine with occipital nerve tenderness. Pain. 2015 Dec;156(12):2585-2594. doi: 10.1097/j.pain.0000000000000373. PMID 26447705
- [Result] Vanelderen P, Rouwette T, De Vooght P, Puylaert M, Heylen R, Vissers K, Van Zundert J. Pulsed radiofrequency for the treatment of occipital neuralgia: a prospective study with 6 months of follow-up. Reg Anesth Pain Med. 2010 Mar-Apr;35(2):148-51. doi: 10.1097/aap.0b013e3181d24713. PMID 20301822
- [Result] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266